CLINICAL TRIAL: NCT04774783
Title: Pilot Study on the Effects of Low-Level Laser Therapy Treatment for Acute and Persistent Discomfort
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arkansas Colleges of Health Education (Other)
Responsible Party: Principal Investigator, Daniel Curtis, Director of Clinical Education, Arkansas Colleges of Health Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT-2020-006
Record Dates: First submitted 2021-02-20; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Chronic Pain; Acute Pain
MeSH Terms: conditions — Chronic Pain; Acute Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Low-Level Laser Therapy (Experimental): Over the course of the study, participants within this group will receive 12 sessions of Low-Level Laser Therapy (LLLT) treatment over a duration of 4 weeks using the Richmar TheraTouch LX2 device. Treatment location will be determined through assessment of each qualifying participant. Treatment sessions will be limited to a single area of the body associated with the qualifying participant's primary pain complaint.
  Interventions: Device: Low-Level Laser Therapy

INTERVENTIONS:
Device: Low-Level Laser Therapy — The TheraTouch LX2 device includes a 9-diode cluster probe which emits a combination of LED and laser light. The cluster probe includes four 650 nm LED diodes capable of delivering a total of 40 mW and five 850 nm laser diodes capable of delivering a total of 1000 mW of power. LLLT will the applied with the cluster probe directly in contact with the subject's skin. LLLT dosages will vary according to the location of the subject's pain and may require multiple applications during a session. Each individual application will typically range from 4-16 Joules.

SUMMARY:
This study will examine the effectiveness of Low-Level Laser Therapy (LLLT) for the management of pain in various locations of the body. All subjects selected for participation in the study will be assigned to a LLLT treatment group for a duration of 12 sessions.

DETAILED DESCRIPTION:
Low-Level Laser Therapy (LLLT) is a treatment modality that is gaining popularity in the field of physical therapy for its proposed mediation of pain. LLLT is typically used in conjunction with other more conventional physical therapy treatment sessions; therefore, it is not clear if the benefits are from the LLLT or the conventional treatment, or the combination of them both. The research question: Does low-level laser therapy treatment with a class 3B Laser decrease pain and improve function in persons with persistent or acute joint/muscle discomfort as compared to before treatment?

Study participants presenting with pain will be interviewed regarding the location and intensity of their primary pain complaints. Participants will also be asked to identify functional limitations associated with their pain. Participants will undergo an initial screening process to identify the presence of any exclusion factors and precautions associated with the delivery of LLLT. Investigators will collect pre-test and post-test information from participants regarding pain intensity and perceived functional limitations. Investigators will also collect relevant joint range of motion and muscle strength data during the first and last sessions. Treatment location for the study will vary within the participant group and will be determined during the initial screening process. The intervention will include LLLT treatment using a combination of LED and laser light delivered by the Richmar TheraTouch LX2 device.

ELIGIBILITY:
Inclusion Criteria:

* subjects having persistent or acute discomfort/pain in a muscle or joint of their body
* ability to speak English or provide own translator
* ability to complete the pre-test/post-test session
* ability to attend three times per week

Exclusion Criteria:

* pregnant women
* currently undergoing immunosuppression therapy
* subjects with photosensitivity concerns

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-03-26 (Estimated); Study Completion 2021-03-26 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Visit 1, Week 1 of 4
  The NPRS is an eleven point scale (0-10) where the subject is asked to provide a rating of their pain current, best and worst pain intensity over the past 24 hours. Subjects are asked to rate their pain on a scale of 0 to 10 with 0 being "No Pain" and 10 being "Worst Pain Imaginable". Data will be collected at baseline during Visit 1.
Numeric Pain Rating Scale (NPRS) | Visit 12, Week 4 of 4
  The NPRS is an eleven point scale (0-10) where the subject is asked to provide a rating of their pain current, best and worst pain intensity over the past 24 hours. Subjects are asked to rate their pain on a scale of 0 to 10 with 0 being "No Pain" and 10 being "Worst Pain Imaginable". Data will be collected post-treatment during Visit 12.
Patient-Specific Functional Scale (PSFS) | Visit 1, Week 1 of 4
  The PSFS is a device used to quantify the extent of a subject's perceived functional limitations due to a particular problem or condition. The subject is asked to identify up to three activities in which they feel their performance is limited. For each of the activities identified, the subject will rate their perceived level of limitation using an eleven point scale (0-10) with 0 being "Unable to perform activity" and 10 being "Able to perform activity at the same level as before injury or problem". Data will be collected at baseline during Visit 1.
Patient-Specific Functional Scale (PSFS) | Visit 12, Week 4 of 4
  The PSFS is a device used to quantify the extent of a subject's perceived functional limitations due to a particular problem or condition. The subject is asked to identify up to three activities in which they feel their performance is limited. For each of the activities identified, the subject will rate their perceived level of limitation using an eleven point scale (0-10) with 0 being "Unable to perform activity" and 10 being "Able to perform activity at the same level as before injury or problem". Data will be collected post-treatment during Visit 12.
Joint Range of Motion | Visit 1, Week 1 of 4
  Relevant range of motion data will be collected from each qualifying subject at baseline during Visit 1.
Joint Range of Motion | Visit 12, Week 4 of 4
  Relevant range of motion data will be collected from each qualifying subject post-treatment during Visit 12.
Muscle Strength | Visit 1, Week 1 of 4
  Relevant muscle strength data will be collected from each qualifying subject via manual muscle test or dynamometer at baseline during Visit 1.
Muscle Strength | Visit 12, Week 4 of 4
  Relevant muscle strength data will be collected from each qualifying subject via manual muscle test or dynamometer post-treatment during Visit 12.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Curtis, DPT, Principal Investigator — Arkansas Colleges of Health Education
Locations (1):
- Arkansas Colleges of Health Education, Fort Smith, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No